CLINICAL TRIAL: NCT05472909
Title: Music Interventions During Wide-Awake Hand Surgery: A Randomized Controlled Trial
Brief Title: Music Interventions During Wide-Awake Hand Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2022-0674; Protocol Version 4/7/2023 (Other: UW Madison); A536100 (Other: UW Madison)
Record Dates: First submitted 2022-07-21; First posted 2022-07-25 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2025-10

CONDITIONS: Anxiety; Surgery
Keywords: wide-awake hand surgery; music intervention; patient care
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standardized Relaxation Music (Experimental)
  Interventions: Other: Standardized Relaxation Music
- Personal Choice of Music (Active Comparator)
  Interventions: Other: Personal Choice of Music

INTERVENTIONS:
Other: Standardized Relaxation Music — Participants listen to standardized relaxation music during surgery.
  Arms: Standardized Relaxation Music
Other: Personal Choice of Music — Participants listen to their preferred music during surgery.
  Arms: Personal Choice of Music

SUMMARY:
The purpose of this study is to examine if patients have a lower anxiety level during wide awake hand surgery while listening to their choice of music vs standardized relaxation music. Patients who are planning to undergo wide awake (local anesthetic only hand surgery) and agree to participate will be randomized to either a music intervention where they listen to their choice of music genre or standardized relaxation music during their time in the operating room. 170 participants will be enrolled and can expect to be on study for 2 weeks.

DETAILED DESCRIPTION:
Music has been shown to decrease anxiety and pain during surgery. Wide awake local anesthesia no tourniquet (WALANT) surgery on the hand is gaining popularity due to efficiency, cost savings and patient safety.

Despite the popularity of WALANT, it still can be anxiety producing even for patients who choose to proceed with surgery without sedation. Music has been shown to decrease anxiety during surgery, but patients' music choices vary widely. The frequency (Hz) of the music intervention has been shown to impact pain reduction, and patient choice of music has been shown to increase sense of control which can decrease anxiety. No study has evaluated the intraoperative effect of patient choice of music vs standardized relaxation music on intraoperative anxiety.

The primary objective of this research is to compare the effect of patient music choice vs standardized relaxation music played during surgery on anxiety levels in patients undergoing WALANT hand surgery. The investigators hypothesize that standardized relaxation music will result in reduced anxiety compared to patient's choice of music.

ELIGIBILITY:
Inclusion Criteria:

* Adult (18 years of age or older) patients
* Undergoing Wide Awake Local Anesthesia No Tourniquet (WALANT) hand surgery

Exclusion Criteria:

* Patients under the age of 18
* Patients unable to consent for themselves
* Patients unwilling to consent
* Non-English speaking patients
* Patients with significant hearing impairment not able to be corrected with assistive devices

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Change in Visual Analog Scale-Anxiety (VAS-A) Score | day 0 post-operative, up to day 14
  The VAS-A is scored from 0-10 where 0 is 'feeling calm' and 10 is 'extremely anxious'.
Change in State Trait Anxiety Inventory (STAI) Score | day 0 post-operative, up to day 14
  The STAI is a 20-item questionnaire (form Y-1) scored on a 4 point likert scale where 1 is 'not at all', 2 is 'somewhat', 3 is 'moderately so', and 4 is 'very much so' for a total possible range of scores from 20-80 where higher scores indicate increased anxiety.

SECONDARY OUTCOMES:
Participant Heart Rate | day 0, pre- and intraoperative
Participant Systolic Blood Pressure | pre- and intraoperative on day 0
Participant Diastolic Blood Pressure | pre- and intraoperative on day 0
Participant Respiratory Rate | pre- and intraoperative on day 0

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Kruse, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No
Results will not be shared with patients or their primary care physicians. Study results will be shared via manuscript publication in a peer reviewed journal. Data will be pooled and deidentified. No individual results will be shared.

REFERENCES:
- [Background] Kuhlmann AYR, de Rooij A, Kroese LF, van Dijk M, Hunink MGM, Jeekel J. Meta-analysis evaluating music interventions for anxiety and pain in surgery. Br J Surg. 2018 Jun;105(7):773-783. doi: 10.1002/bjs.10853. Epub 2018 Apr 17. PMID 29665028
- [Background] Palmer JB, Lane D, Mayo D, Schluchter M, Leeming R. Effects of Music Therapy on Anesthesia Requirements and Anxiety in Women Undergoing Ambulatory Breast Surgery for Cancer Diagnosis and Treatment: A Randomized Controlled Trial. J Clin Oncol. 2015 Oct 1;33(28):3162-8. doi: 10.1200/JCO.2014.59.6049. Epub 2015 Aug 17. PMID 26282640
- [Background] Bradt J, Dileo C, Shim M. Music interventions for preoperative anxiety. Cochrane Database Syst Rev. 2013 Jun 6;2013(6):CD006908. doi: 10.1002/14651858.CD006908.pub2. PMID 23740695
- [Background] Feneberg AC, Kappert MB, Maidhof RM, Doering BK, Olbrich D, Nater UM. Efficacy, Treatment Characteristics, and Biopsychological Mechanisms of Music-Listening Interventions in Reducing Pain (MINTREP): Study Protocol of a Three-Armed Pilot Randomized Controlled Trial. Front Psychiatry. 2020 Nov 4;11:518316. doi: 10.3389/fpsyt.2020.518316. eCollection 2020. PMID 33329075
- [Background] Mitchell LA, MacDonald RA. An experimental investigation of the effects of preferred and relaxing music listening on pain perception. J Music Ther. 2006 Winter;43(4):295-316. doi: 10.1093/jmt/43.4.295. PMID 17348757